CLINICAL TRIAL: NCT07029776
Title: A Phase 2 Study Exploring the Use of Bispecific Antibodies to Improve Progression Free Survival in Patients With High-Risk Newly Diagnosed Multiple Myeloma (MMulti-Immune HR)
Brief Title: MMulti-Immune HR; Multi-Target Immunotherapy for High-Risk Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 297250; 64407564MMY201 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2025-05-23; First posted 2025-06-19 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma (MM)
Keywords: Bispecific Antibodies; High-Risk Newly Diagnosed Multiple Myeloma; Multi-Target Immunotherapy; High-Risk Multiple Myeloma; Teclistamab; Daratumumab
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Maintenance; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MRD-negative (Experimental): Subjects who are MRD-negative (a threshold of 10^5) will be given teclistamab+daratumumab followed by talquetamab+daratumumab each for 4 cycles followed by 2-year fixed duration treatment with daratumumab and lenalidomide extended/maintenance therapy for a maximum of 24 cycles, or until myeloma progression.
  Interventions: Drug: teclistamab+daratumumab followed by talquetamab+daratumumab followed by duration treatment with daratumumab and lenalidomide extended/maintenance
- MRD-positive (Experimental): Subjects who are MRD-positive (a threshold of 10^5) will receive a single melphalan (MEL)-based hematopietic stem cell transplantation (HSCT) followed by teclistamab+daratumumab followed by talquetamab+daratumumab each for 4 cycles followed by a 2-year fixed duration treatment with daratumumab and lenalidomide extended/maintenance therapy for a maximum of 24 cycles, or until myeloma progression. MRD status with classification threshold of 10^5 will be assessed by standardized flow cytometry.
  Interventions: Procedure: melphalan (MEL)-based hematopietic stem cell transplantation (HSCT) followed by drug therapy

INTERVENTIONS:
Drug: teclistamab+daratumumab followed by talquetamab+daratumumab followed by duration treatment with daratumumab and lenalidomide extended/maintenance — teclistamab+daratumumab followed by talquetamab+daratumumab each for 4 cycles followed by 2-year fixed duration treatment with daratumumab and lenalidomide extended/maintenance therapy for a maximum of 24 cycles, or until myeloma progression.
  Other Names: JNJ-64407564; Anti-GPRC5D × CD3 Antibody; Talvey; JNJ-54767414; Darzalex; JNJ-64007957; Tecvayli
  Arms: MRD-negative
Procedure: melphalan (MEL)-based hematopietic stem cell transplantation (HSCT) followed by drug therapy — Subjects who are MRD-positive (a threshold of 10^5) will receive a single melphalan (MEL)-based hematopietic stem cell transplantation (HSCT) followed by teclistamab+daratumumab followed by talquetamab+daratumumab each for 4 cycles followed by a 2-year fixed duration treatment with daratumumab and lenalidomide extended/maintenance therapy for a maximum of 24 cycles, or until myeloma progression.
  Arms: MRD-positive

SUMMARY:
The purpose of this research is to learn whether using teclistamab and talquetamab at different time points will improve survival in participants with high-risk Multiple Myeloma (MM).

The treatment on this study will consist of Induction chemotherapy and stem cell collection, Immunotherapy 1 chemotherapy and Immunotherapy 2 chemotherapy. For participants whose testing show they are Minimal Residual Disease (MRD) positive (still have myeloma cells present in the bone marrow testing), a Melphalan-based stem cell transplant will be performed. For participants whose testing show they are MRD negative, the stem cell transplant will not be performed. All participants will go on to receive Immunotherapy 3 chemotherapy, Immunotherapy 4 chemotherapy, and Maintenance therapy.

DETAILED DESCRIPTION:
The two primary objectives are to determine (1) the Complete Response Rate (CRR) and (2) the 2-year Progression-Free Survival (PFS) percentage in participants with high-risk multiple myeloma (HRMM) treated with the sequential use of Bispecific Antibodies.

Overview of Study Design:

We will implement a Phase 2 clinical trial to explore the use of early and late bispecific antibodies consolidation and extended/maintenance therapy as a way of overcoming intraclonal heterogeneity and improving PFS in HRMM. Subjects will receive induction treatment with daratumumab (Dara)-KRD for 4 cycles to obtain immediate disease control, reduce tumor bulk and minimize the risk of subsequent cytokine release syndrome (CRS). Peripheral blood stem cell (PBSC) will be harvested after induction treatment. Immune therapy will consist of teclistamab+daratumumab followed sequentially by talquetamab+daratumumab each for 4 cycles. Next, an MRD-based consolidation approach will be utilized where subjects who are MRD-negative (a threshold of 10^5) will be given teclistamab+daratumumab followed by talquetamab+daratumumab each for 4 cycles followed by 2-year fixed duration treatment with daratumumab and lenalidomide extended/maintenance therapy for a maximum of 24 cycles, or until myeloma progression. Subjects who are MRD-positive (a threshold of 10^5) will receive a single melphalan (MEL)-based hematopietic stem cell transplantation (HSCT) followed by teclistamab+daratumumab followed by talquetamab+daratumumab each for 4 cycles followed by a 2-year fixed duration treatment with daratumumab and lenalidomide extended/maintenance therapy for a maximum of 24 cycles, or until myeloma progression. Minimal residual disease (MRD) status with classification threshold of 10^5 will be assessed by standardized flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed active MM requiring treatment. Patients with a previous history of smoldering myeloma will be eligible if there is evidence of PD requiring initiation of treatment.
* Patients must be either untreated or have not received more than two months of MM therapy. However, bisphosphonates and localized radiation are allowed.
* Patients must have clinical features of high-risk disease, at time of initial diagnosis or initial assessment prior to enrollment, which may include one or more of the following:

  * High-risk cytogenetic abnormalities, including t(4;14), t(14;16), t(14;20), del17p13, del1p, or gain 1q with del1p by FISH, with a cutoff point of 20% or greater.
  * Beta-2-microglobulin >5.5 mg/L with normal kidney function test per the institutional reference.
  * Presence of extramedullary disease defined as soft tissue plasmacytoma (excluding Paramedullary/Paraskeletal plasmacytoma)
  * ≥ 3 focal lesions on F18-fluorodeoxyglucose positron emission tomography (FDG-PET) imaging
  * LDH ≥ 360 U/L (Rule out hemolysis and infection; contact Principal Investigator if any doubt.)
  * Circulating plasma cells ≥5 percent of white blood cells on conventional peripheral blood smear (manual white blood cell differential count) or peripheral blood flow cytometry.
* ECOG ≤ 2, unless solely due to symptoms of MM-related bone disease.
* Patients must have a platelet count ≥ 50,000/μL and hemoglobin level of ≥7.5 g/dl and absolute neutrophilic count (ANC) of 1.0x10^9/L unless lower levels are explained by extensive BM plasmacytosis.
* Patients must be at least 18 years of age and not older than 75 years of age at the time of consent.
* Patients must have adequate renal function with baseline serum creatinine level < 3 mg/dL and estimated creatinine clearance ≥30 mL/min. Creatinine clearance may be calculated using Cockcroft-Gault, eGFR (MDRD), or CKD-epi formula and baseline Alanine Aminotransferase (ALT) < 3x Upper Limit of Normal (ULN).
* Patients must have an ejection fraction by echocardiogram (ECHO) or Multigated Acquisition (MUGA) scan ≥ 45%
* Patients must have adequate pulmonary function studies > 50% of predicted on mechanical aspects (FEV1, FVC, etc.) and diffusion capacity (DLCO) > 50% of predicted. If the patient is unable to complete pulmonary function tests (PFT) due to MM related pain or other conditions, an exception may be granted if the Principal Investigator documents that the patient is a candidate for high dose therapy.
* Patients must have signed an IRB-approved informed consent form (ICF) indicating their understanding of the proposed treatment and that the protocol has been approved by the IRB.
* Female subjects must use effective methods of birth control during the course of the study and for 6 months after stopping study medications.
* Female subjects must not donate eggs during the study and for 6 months after the last dose of study medications.
* Male subjects must not donate sperm during the study and for 3 months after the last dose of study medications.

Exclusion Criteria:

* Poorly controlled hypertension, diabetes mellitus, or other serious medical or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol.
* Patients must not have prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, low Gleason score prostate cancer on active surveillance or having had surgery/radiation with curative intent within one year of consent or other cancer for which the patient has not received treatment for one year prior to consent. Other cancers will only be acceptable if the patient's life expectancy exceeds five years.
* Pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 3 months after the last dose of any component of the treatment regimen. Or subject is a man who plans to father a child while enrolled in this study or within 3 months after the last dose of any component of the treatment regimen. Women of childbearing potential (WOCBP) must have a negative pregnancy documented within one week of consent. Subjects of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal. Note that FEV1 testing is required for subjects suspected of having COPD and patients must be excluded if FEV1 is <50% of predicted normal.
* Moderate or severe persistent asthma within the past 2 years, or uncontrolled asthma of any classification. Note that patients who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate in the study.
* Active autoimmune disease
* Active systematic viral, fungal or bacterial infection, requiring systemic therapy.
* Clinically significant cardiac disease, including Myocardial infarction within 6 months before consent, or Uncontrolled cardiac arrhythmia or unstable or uncontrolled disease/condition related to or affection cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class 3-4) (Appendix 1)
* Patient is:

  * seropositive for human immunodeficiency virus (HIV)
  * seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]. Subjects with resolved infection (i.e., subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs] must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) levels. Those with active infection will be excluded. Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) and a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
  * Seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).
* Patients who received plasmapheresis within 28 days of start of study treatment at Induction with Dara-KRD.
* Patients with focal radiation therapy within 14 days prior to consent with the exception of palliative radiotherapy for symptomatic management but not on measurable extramedullary plasmacytoma.
* Known history of allergy to Captisol ® (a cyclodextrin derivative used to solubilize carfilzomib).
* Known history of allergy, hypersensitivity, or intolerance to boron or mannitol, sorbitol, corticosteroids, monoclonal antibodies or human proteins, or their excipients.
* Known intolerance or allergy to lenalidomide.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-04-01 (Estimated); Study Completion 2032-04-01 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate (CRR) in subjects with high-risk multiple myeloma (HRMM) treated with the sequential use of Bispecific Antibodies. | Up to 4 years
  to determine the Complete Response Rate (CRR), defined as the proportion of subjects achieving complete response (CR) or stringent complete response (sCR) according to IMWG criteria at the 'Pre-Maintenance' timepoint (after completion of Immunotherapy #4, Cycle 4)
the 2-year Progression-Free Survival (PFS) percentage in subjects with high-risk multiple myeloma (HRMM) treated with the sequential use of Bispecific Antibodies. | 2 years after study completion
  determine the 2-year Progression-Free Survival (PFS) percentage in subjects with high-risk multiple myeloma (HRMM) treated with the sequential use of bispecific antibodies.

SECONDARY OUTCOMES:
evaluate the Minimal Residual Disease (MRD) Negativity Rate (MRDNR) in subjects with HRMM treated with the sequential use of Bispecific Antibodies. | Up to 4 years
  to evaluate the Minimal Residual Disease (MRD) Negativity Rate (MRDNR) in subjects with high-risk multiple myeloma (HRMM) treated with the sequential use of bispecific antibodies. MRDNR will be determined using FDA-approved clonoSEQ NGS assessment at a threshold of 10^6.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No